CLINICAL TRIAL: NCT05148884
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Preliminary Efficacy of NLX-112 Versus Placebo in Levodopa-induced Dyskinesia in Parkinson's Disease
Brief Title: Study to Assess the Safety, Tolerability and Preliminary Efficacy of NLX-112 Versus Placebo in L-dopa-induced Dyskinesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurolixis SAS (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); Parkinson's UK (Other); CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NLX-112-DYS-101
Record Dates: First submitted 2021-10-07; First posted 2021-12-08 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Medication-Induced Dyskinesia
Keywords: Levodopa; Dyskinesia; Parkinson´s disease; L-dopa; NLX-112; Befiradol; LID
MeSH Terms: conditions — Dyskinesia, Drug-Induced; Dyskinesias; Parkinson Disease | interventions — befiradol; PHA-568487E

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled Phase 2a study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NLX-112 (Experimental): Patients will self-administer NLX-112 2 times each day, once in the morning and once in the evening. Up-titration over 4 weeks, maximal dose of 2 mg/day during 2 weeks, down-titration over 2 weeks.
  Interventions: Drug: NLX-112
- Placebo (Placebo Comparator): Patients will self-administer placebo 2 times each day, once in the morning and once in the evening. Up-titration of number of tablets over 4 weeks, number of tablets equivalent to maximal dose of 2 mg/day NLX-112 during 2 weeks, down-titration over 2 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NLX-112 — NLX-112 will be supplied as tablets containing 0.25 mg NLX-112. NLX-112 is a structurally novel centrally acting, high-efficacy selective 5-HT1A receptor agonist with nanomolar affinity for 5-HT1A receptors. Proposed as a treatment for L-DOPA-induced-dyskinesia in Parkinson's disease.
  Other Names: F13640; befiradol; 4-piperidinemethanamine; 1-(3-chloro-4-fluorobenzoyl)-4-fluoro-N-[(5-methyl-2-pyridinyl)-methyl]; (2E)-2-butenedioate
  Arms: NLX-112
Drug: Placebo — Placebo will be matching tablets (identical weight, shape and color) without NLX-112.
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled Phase 2a study evaluating the safety, tolerability, and preliminary efficacy of up to 2 mg/day (1 mg BID) of NLX-112 versus placebo in patients with moderate to severe L-DOPA induced dyskinesia (LID) in Parkinson's disease (PD). NLX-112 will be up-titrated to either 2 mg/day or to the highest well-tolerated dose less than 2 mg/day over 4 weeks, maintained at the well-tolerated dose for an additional 2 weeks, and then down-titrated over 2 weeks.

DETAILED DESCRIPTION:
This is a two-arm, double-blind, randomized, placebo-controlled Phase 2a study evaluating the safety, tolerability, and preliminary efficacy of up to 2 mg/day of NLX 112 versus placebo in patients with moderate to severe L-DOPA induced dyskinesia (LID) in Parkinson's disease (PD). NLX-112 will be up-titrated to either 2 mg/day (1 mg BID) or to the highest well-tolerated dose less than 2 mg/day over 4 weeks, maintained at the well-tolerated dose for an additional 2 weeks, and then down-titrated over 2 weeks.

Patients will report to the study clinic for a screening visit (Visit 1), followed by a baseline visit on Day 1 (Visit 2) where patients will be randomized and begin treatment. Two remote safety visits over telephone (Days 7 and 49 [Visit 3 and Visit 8]) will be conducted. Once treatment has commenced, there will be 2 in-person safety visits to the clinic (Days 14 and 21 [Visit 4 and Visit 5]), 2 in-person efficacy visits to the clinic (Days 28 and 42 [Visit 6 and Visit 7]) and one follow-up in person final safety visit (Day 70 [Visit 9]). In total, patients will report to the clinic for 7 in-person visits. Patients entering the study will be randomized in a 2:1 ratio (16:8 patients) to receive either NLX 112 or placebo.

At Visits 2, 6 and 7, efficacy assessments will start 30 minutes after the patient has taken 150% of his or her regular L-DOPA dose, when the patient is ON and experiencing typical dyskinesia.

A PD Home Dyskinesia Diary (electronic) will be completed by the patients and/or caregiver with concordance in ON time with dyskinesia between study staff and patient. Two consecutive 24-hour diaries will be completed prior to randomization (baseline, Visit 2) and prior to the clinic visits on Days 28 and 42 (Visits 6 and 7).

A wearable dyskinesia assessment device will be used to monitor dyskinesias during a 2-day period prior to the baseline visit (Day 1, Visit 2) and a 2-day period prior to the clinic visits on Days 28 and 42 (Visits 6 and 7, respectively).

Blood will be collected for possible NLX-112 plasma concentration measurements on Days 14, 21, 28, 42 and 70 (Visits 4, 5, 6, 7 and 9).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 30 - 85 years old (inclusive) with a diagnosis of idiopathic PD according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnosis criteria.
2. PD patient is stably and optimally treated with L-DOPA; other anti-PD treatments are allowed if used for at least 4 weeks of previous continuous treatment.
3. Patient agrees to be challenged with 150% of their normal L-DOPA dose (maximum L-DOPA dose 250 mg) 30 minutes prior to efficacy assessments at baseline (Visit 2) and at the 2 efficacy clinic visits (Visits 6 and 7).
4. PD patient exhibits troublesome peak-dose LID, confirmed by a score of at least 1 on part IV, item 33 (disability) of the UPDRS at screening (Visit 1) and at Day 1 (baseline, Visit 2).
5. At least 90 minutes in total for each 24-hour period during 2 days are indicated as "ON with troublesome dyskinesia" (according to the PD Home Dyskinesia Diary) prior to Day 1 (baseline, Visit 2).
6. Patient (and/or caregiver) demonstrates ability to accurately complete the PD Home Dyskinesia Diary entries during the screening visit.
7. Patient can read well enough to understand the informed consent document and other subject materials.
8. Female patients of child-bearing potential must have a negative urine pregnancy test at screening (Visit 1) and on Day 1 (Visit 2), must agree to avoid pregnancy during the study, and must practice abstinence (only allowed when this is the preferred and usual lifestyle of the subject) or must agree to use a highly effective method of contraception with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD] or intrauterine hormone-releasing system [IUS]) starting from 4 weeks prior to administration of the study drug and continuing during the course of the study until 4 weeks after last after IMP administration. Female subjects must agree to refrain from donating eggs from the date of dosing until 3 months after dosing with the IMP. Their male partner must agree to use a condom during the same time frame if he has not undergone vasectomy.

Females of non-childbearing potential are defined as pre-menopausal females who are sterilised (tubal ligation or permanent bilateral occlusion of fallopian tubes); or females who have undergone hysterectomy or bilateral oophorectomy; or post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with detection of follicle stimulating hormone [FSH] 25-140 IE/L is confirmatory).

Male patients must be either vasectomised, consent to use condom or practice sexual abstinence to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the date of dosing until 3 months after dosing with the IMP. Their female partner of child-bearing potential must use highly effective contraceptive methods with a failure rate of < 1% to prevent pregnancy (see above) during the same period.

Exclusion Criteria:

1. Patient has severe PD with a Hoehn and Yahr stage = 5.
2. Patient has unstable medical status, prior brain surgery against tumors or hemorrhage (excluding deep brain stimulation [DBS], i.e., DBS patients will be allowed to be enrolled) or is scheduled to receive surgery during the trial period.
3. Patient has orthostatic hypotension: a decrease in systolic blood pressure (at least 20 mm Hg) or diastolic blood pressure (at least 10 mm Hg) within 3 minutes of the patient standing up, compared to pressures obtained while in a sitting position for at least 5 minutes. At screening and baseline visits (Visit 1 and Visit 2), vital signs to assess orthostatic hypotension will be conducted in triplicate, 15-20 minutes apart, with the average of the 3 assessments used for exclusion.
4. Patient has dementia (MMSE <20).
5. Patient has clinically significant renal or liver disorder.
6. Patient currently exhibits generalized obsessive-compulsive disorder, panic disorder, bipolar disorder, post-traumatic stress syndrome (PTSD), clinically significant parasomnias or any other psychotic disorder as established by structured clinical interview for DSM disorders (SCID). Visual hallucinations are allowed.
7. Any suicidal actions in the past 2 years (per investigator judgement i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior).
8. Any suicidal ideation of type 4 or 5 in the C-SSRS in the past 3 months (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent).
9. Patient has taken an anti-convulsant, an anti-psychotic (except quetiapine), pindolol, tertatolol or buspirone within 4 weeks of baseline (Day 1, Visit 2).
10. Patient has taken any medication, within 4 weeks of baseline (Day 1, Visit 2) that inhibits or up-regulates CYP4503A4.
11. Patient is concurrently participating in another investigational drug trial or has participated in another investigational drug trial within the past 3 months.
12. Patient is at high risk of non-compliance in the Investigator's opinion.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Newman-Tancredi, PhD, Study Director — Neurolixis SAS; Per Svenningsson, Professor, Principal Investigator — ASC Torsplan
Locations (5):
- Sweden (5):
  - Sahlgrenska Hospital, Gothenburg
  - Skåne University Hospital, Lund
  - ASC Torsplan, Stockholm
  - Karolinska University Hospital, Solna, Stockholm
  - CTC Clinical Trial Consultants AB (CTC), Uppsala

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants in the study were identified according to the routines of the clinical study sites.
  Patients were recruited at 5 clinical sites, with a planned average of 4 to 6 patients per site.
Pre-assignment Details: A total of 35 patients were screened and 27 were randomized and dosed in the study. Eighteen patients were allocated to treatment with NLX-112 and 9 were allocated to placebo. Twenty-three patients, 15 on NLX-112 and 8 on placebo, completed the study.
Groups:
- NLX-112: Patients were randomized to receive either active treatment with NLX-112 or placebo. This arm represents the patients that received NLX-112 oral tablets, uptitrated over 4 weeks to a maximal daily dose of 2 mg for 14 days given as 1mg two times a day.
- Placebo: Patients were randomized to receive either active treatment with NLX-112 or placebo. This arm represents the patients that received placebo.
Period: Overall Study
Arm/Group | NLX-112 | Placebo
Started | 18 | 9
Completed | 15 | 8
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Deep brain stimulation operation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- NLX-112: Patients were randomized to receive either active treatment with NLX-112 or placebo. This arm represents the patients that received NLX-112.
- Total: Total of all reporting groups
Arm/Group | NLX-112 | Placebo | Total
Number analyzed (Participants) | 18 | 9 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 12
  >=65 years | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (9.7) | 64.6 (6.3) | 65.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 17 | 9 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 9 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 18 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of patients with Adverse events (AEs) divided into categories of severity/intensity (grade 1 to grade 5 following the common terminology criteria for AEs (CTCAE) v5.0) and assessed relationship to IMP (unlikely, possibly or probably related). AEs (including SAEs) were collected from the start of IMP administration until the end-of-study visit.
Time Frame: AEs (including SAEs) were collected from the start of IMP administration until the end-of-study visit. Through study completion, an average of 10 weeks.
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 18 | 9
Participants
  Any AE | 16 | 7
  Any SAE | 0 | 1
  Congenital Anomaly or Birth Defect | 0 | 0
  Persistent or Significant Disability/Incapacity | 0 | 0
  Requires or Prolongs Hospitalization | 0 | 1
  Is Life Threatening | 0 | 0
  Other Medically Important Serious Event | 0 | 0
  Any AE leading to withdrawal from study | 1 | 0
  Any AE leading to death | 0 | 0
  Causality - Unlikely Related | 11 | 4
  Causality - Possibly Related | 15 | 5
  Causality - Probably Related | 3 | 3
  Action taken with study drug - Dose Not Changed | 12 | 6
  Action taken with study drug - Dose Reduced | 4 | 3
  Action taken with study drug - Drug Interrupted | 0 | 1
  Action taken with study drug - Not Applicable | 5 | 2
  Severity - Mild | 14 | 7
  Severity - Moderate | 10 | 4
  Severity - Severe | 0 | 1
  Severity - Life-Threatening | 0 | 0
  Severity - Death | 0 | 0

2. Primary Outcome: Number of Participants With Any Clinically Significant Changes From Baseline in Electrocardiogram (ECG)
Description: Number of patients with clinically significant changes from baseline in Electrocardiogram (Rate, PR interval, QRS duration, QT, QTcB, and QTcF). Any abnormalities were specified and documented as either clinically significant or not clinically significant.
Time Frame: Visit 1 (Screening), Visit 2 (Baseline, Day 1), Visit 4 (Clinic Safety Visit, Day 14), Visit 5 (Clinic Safety Visit, Day 21), Visit 6 (Clinic Efficacy Visit, Day 28), Visit 7 (Clinic Efficacy Visit, Day 42) and Visit 9 (Follow-up Clinic Visit, Day 70).
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 18 | 9
Participants | 0 | 0

3. Primary Outcome: Number of Patients With Any Clinically Significant Changes From Baseline in Vital Signs
Description: Number of patients with clinically significant changes from baseline in vital signs (Systolic blood pressure (mmHg), diastolic blood pressure (mmHg), Heart rate, respiratory rate, body temperature). Any vital signs outside the normal ranges at each site were judged as either not clinically significant or clinically significant by the clinician.
Time Frame: as for outcome 2
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 18 | 9
Participants | 2 | 0

4. Primary Outcome: Number of Patients With Any Clinically Significant Changes From Baseline in Safety Laboratory Parameters
Description: Number of patients with clinically significant changes from baseline in safety laboratory parameters. Any lab values outside the normal ranges at each site were judged as not clinically significant or clinically significant.
Time Frame: as for outcome 2
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 18 | 9
Participants | 2 | 1

5. Primary Outcome: Number of Patients With Clinically Significant Abnormalities in Physical Examinations
Description: Number of patients with clinically significant abnormalities in physical examination investigated by general appearance, head, ears, eyes, nose, throat, neck, skin, cardiovascular system, respiratory system, abdominal system, and nervous system. Any abnormalities were specified and documented as either clinically significant or not clinically significant.
Time Frame: Visit 1 (Screening) and Visit 9 (Follow-up Clinic Visit, Day 70).
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 18 | 9
Participants
  Visit 1 | 8 | 1
  Visit 9 | 7 | 4

6. Primary Outcome: Number of Patients With Suicidal Ideation/Behavior as Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Number of patients with change from baseline in suicidal ideation/behavior as assessed by C-SSRS questionnaire with no total score summation. The scale contains 6 "yes" or "no" questions in which respondents were asked to indicate whether they have experienced several thoughts or feelings relating to suicide over the past 3 months and behavior over their lifetime using a baseline scale at visit 1 and any cahnges since last visit using a follow-up scale at subsequent visits. Each question addresses a different component of the respondent's suicide ideation severity and behavior. Q1: wish to be dead, Q2: non-specific suicidal thoughts, Q3-5: more specific suicidal thoughts and intent to act, Q6: suicidal behavior over the respondent's lifetime and past 3 months or since last visit for visits after the visit 1.
Time Frame: The baseline scale was used at screening (Visit 1) and the follow-up scale at all subsequent visits (Visit 2, 4-7, 9)
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 18 | 9
Participants | 0 | 0

7. Secondary Outcome: Change From Baseline at the Final Efficacy Clinic Visit (Day 42), After a 150% L-dopa Dose Challenge, in the Unified Dyskinesia Rating Scale (UDysRS) Total Score - Change From Baseline
Description: The Unified Dyskinesia Rating Scale (UDysRS) is a rating instrument designed to assess the core features of dyskinesia in Parkinson´s Disease. The UDysRS consists of 4 parts:
  * Part 1, historical disability with regard to the patient's perceptions of the impact on activities of daily living (ADL) of on-dyskinesia (11 items).
  * Part 2, historical disability with regard to the patient's perceptions of the impact on ADL of off-dystonia (4 items).
  * Part 3, objective impairment, which assesses severity of dyskinesia, affected body parts, and type of impairment (choreic vs. dystonic) (7items).
  * Part 4, objective disability, based on an evaluation of Part 3 activities (4 items).
  Each item in the UDysRS was scored from 0 to 4, with a possible maximum total score sum of 104 where a higher score indicates a worse outcome.
  The UDysRS Parts 3 and 4 were repeated 3 times after each L-dopa challenge, and the timepoint with the worst outcome was used to calculate total score sum
Time Frame: At baseline (Day 1, Visit 2), and Day 42 (Visits 7)
Population: Per protocol analysis set (one patient excluded in placebo arm due to major protocol deviation).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 15 | 7
score on a scale
  Visit 2 Baseline | 31.6 (9.7) | 39.9 (14.2)
  Visit 7 Clinic Efficacy Visit | 25.3 (10.2) | 37.4 (12.8)
Statistical Analysis 1: Comparison: NLX-112; Linear mixed model (LMM) of change from baseline with treatment, visit and the interaction treatment*visit as fixed categorical effects and subject within treatment as a random effect. The baseline value of the dependent variable has been included in the model as a continuous covariate. Kenward-Roger's improved approximation for degrees of freedom (2009) has been used; Test type: Other; p = 0.0016, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.6886, Mixed Models Analysis

8. Secondary Outcome: Change From Baseline in UDysRS Total Score at Day 28, After a 150% L-DOPA Dose Challenge - Change From Baseline
Description: as for outcome 7
Time Frame: At baseline (Day 1, Visit 2) and Day 28 (Visits 6)
Population: Per protocol analysis set (one patient excluded in placebo arm due to major protocol deviation).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 15 | 7
score on a scale
  Visit 2 Baseline | 31.6 (9.7) | 39.9 (14.2)
  Visit 6 Clinic Efficacy Visit | 27.5 (11.2) | 37.9 (14.5)
Statistical Analysis 1: Comparison: NLX-112; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0281, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.7953, Mixed Models Analysis

9. Secondary Outcome: Change From Baseline in Total Objective Score (Parts 3, 4) of the UDysRS at Day 28 and Day 42, After a 150% L-DOPA Dose Challenge - Change From Baseline
Description: The Unified Dyskinesia Rating Scale (UDysRS) is a rating instrument designed to assess the core features of dyskinesia in Parkinson´s Disease. The UDysRS consists of 4 parts:
  * Part 1, historical disability with regard to the patient's perceptions of the impact on activities of daily living (ADL) of on-dyskinesia (11 items).
  * Part 2, historical disability with regard to the patient's perceptions of the impact on ADL of off-dystonia (4 items).
  * Part 3, objective impairment, which assesses severity of dyskinesia, affected body parts, and type of impairment (choreic vs. dystonic) (7items).
  * Part 4, objective disability, based on an evaluation of Part 3 activities (4 items).
  Each item in the UDysRS was scored from 0 to 4, with a possible total score sum for parts 3 and 4 of 44, where a higher score indicates a worse outcome.
  The UDysRS Parts 3 and 4 were repeated 3 times after each levodopa challenge, and the timepoint with the worst outcome was used to calculate total score sum.
Time Frame: At baseline (Day 1, Visit 2), Day 28 and Day 42 (Visits 6 and 7)
Population: Per protocol analysis set (one patient excluded in placebo arm due to major protocol deviation).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 15 | 7
score on a scale
  Visit 2 Baseline | 15.5 (6.2) | 18.1 (7.9)
  Visit 6 Clinic Efficacy Visit | 13.8 (8.5) | 17.1 (7.2)
  Visit 7 Clinic Efficacy Visit | 12.4 (7.2) | 18.0 (7.7)

10. Secondary Outcome: Change From Baseline in ON Time Without Troublesome Dyskinesia (ON Without Dyskinesia Plus ON With Non-troublesome Dyskinesia) Based on a PD Home Dyskinesia Diary - Change From Baseline
Description: A PD Home Dyskinesia Diary (electronic) as completed by the patient and/or caregiver with concordance in ON time with dyskinesia between study staff and patient. The diary was integrated in the Kinesia 360 wearable dyskinesia assessment system and was based on the PD Home Diary developed by Hauser et al 2004. The diary was used to score 5 different conditions in 30-minute time intervals during 2x24 hours prior to Visit 2 (Baseline), Visit 6 (Titration) and Visit 7 (Steady state):
  * ASLEEP;
  * OFF;
  * ON (i.e., adequate control of PD symptoms) without dyskinesia;
  * ON with non-troublesome dyskinesia;
  * ON with troublesome dyskinesia.
  Presented as the ratio of ON Time without troublesome dyskinesia (the sum of the time in ON without dyskinesia together with the time in ON with non-troublesome dyskinesia) compared with the total awake time (ON and OFF).
Time Frame: Baseline - prior to Day 1 (Visit 2), Titration - prior to Day 28 (Visit 6), and Steady state prior to Day 42 (Visit 7).
Population: Per protocol analysis set (one patient excluded in placebo arm due to major protocol deviation).
Measure: Mean (Standard Deviation); unit: Ratio time
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 15 | 7
Ratio time
  Baseline | 0.576 (0.199) | 0.548 (0.192)
  Titration: number analyzed (Participants) | 13 | 6
  Titration | 0.633 (0.133) | 0.591 (0.208)
  Steady-State: number analyzed (Participants) | 12 | 6
  Steady-State | 0.648 (0.182) | 0.564 (0.206)

11. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Scores (Part III, Motor Examination) - Change From Baseline
Description: The UPDRS is one of the most widely-used rating scales employed in the assessment of PD. The UPDRS consists of 4 parts:
  * Part I assesses non-motor experiences of daily living, such as cognitive impairment and depressed mood (4 items).
  * Part II assesses motor experiences of daily living, such as speech and eating tasks (13 items).
  * Part III is a motor examination conducted by the clinician, including assessments of symptoms such as rigidity and tremor (27 items).
  * Part IV is an assessment of motor complications, such as time spent with dyskinesia and functional impact of dyskinesias (11 items).
  Each item in the UPDRS was scored from 0 to 4 (7 items in Part IV was scored 0 to 1), and the individual scores were summed to give a total score that indicates the severity of the disease, with a score of 0 indicating no disability and a score of 199 being the most severe (indicating total disability). Total score sum for Part III alone is 108.
Time Frame: At baseline (Day 1, Visit 2), Day 28 (Visit 6), Day 42 (Visit 7) and Day 70 (Visit 9).
Population: Per protocol analysis set (one patient excluded in placebo arm due to major protocol deviation).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 15 | 7
score on a scale
  Visit 2 Baseline | 17.5 (9.4) | 17.0 (10.3)
  Visit 6 Clinic Efficacy Visit | 13.9 (8.8) | 18.3 (11.5)
  Visit 7 Clinic Efficacy Visit | 13.9 (8.5) | 17.1 (10.5)
  Visit 9 Follow-up Clinic Visit | 14.8 (8.1) | 14.6 (9.0)

12. Secondary Outcome: Change From Baseline in UPDRS Combined Scores (Parts I, II, III and IV) - Change From Baseline
Description: The UPDRS is one of the most widely-used rating scales employed in the assessment of PD. The UPDRS consists of 4 parts:
  Part I assesses non-motor experiences of daily living, such as cognitive impairment and depressed mood (4 items).
  Part II assesses motor experiences of daily living, such as speech and eating tasks (13 items).
  Part III is a motor examination conducted by the clinician, including assessments of symptoms such as rigidity and tremor (27 items).
  Part IV is an assessment of motor complications, such as time spent with dyskinesia and functional impact of dyskinesias (11 items).
  Each item in the UPDRS was scored from 0 to 4 (7 items in Part IV was scored 0 to 1), and the individual scores were summed to give a total score that indicates the severity of the disease, with a score of 0 indicating no disability and a score of 199 being the most severe (indicating total disability).
Time Frame: At baseline (Day 1, Visit 2), Day 28 (Visit 6), Day 42 (Visit 7) and Day 70 (Visit 9).
Population: Per protocol analysis set (one patient excluded in placebo arm due to major protocol deviation).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 15 | 7
score on a scale
  Visit 2 Baseline | 37.0 (13.3) | 41.3 (15.0)
  Visit 6 Clinic Efficacy Visit | 30.5 (13.1) | 37.7 (12.5)
  Visit 7 Clinic Efficacy Visit | 31.3 (13.9) | 37.4 (12.7)
  Visit 9 Follow-up Clinic Visit | 32.6 (12.5) | 34.0 (14.3)

13. Secondary Outcome: Number of Patients in Each Category of Clinical Global Impression of Change (CGI-C) in Overall PD Symptoms
Description: The CGI-C is a clinician-oriented scale that assesses the total improvement in the patient's condition relative to the clinical global impression of severity (CGI-S) scale conducted at baseline.
  1 - Normal not ill, 2 - Borderline ill, 3 - Mildly ill, 4 - Moderately ill, 5 - Markedly ill, 6- Severely ill, 7 - Among the most extremely ill patients The CGI-C rates the patient's condition from 1 to 7: 1 - Very much improved, 2 - Much improved, 3 - Minimally improved, 4 - No change, 5 - Minimally worse, 6 - Much worse, 7 - Very much worse
Time Frame: Clinician rated the patient´s global condition using CGI-S at baseline (Day 1, Visit 2) and CGI-C at Day 28 (Visit 6) and Day 42 (Visit 7).
Population: Per protocol analysis set (one patient excluded in placebo arm due to major protocol deviation).
Measure: Count of Participants; unit: Participants
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 15 | 7
Participants
  Visit 2 Baseline - Normal, not at all ill | 3 | 2
  Visit 2 Baseline - Moderately ill | 8 | 2
  Visit 2 Baseline - Markedly ill | 3 | 2
  Visit 2 Baseline - Severely ill | 1 | 1
  Visit 6 Clinic Efficacy Visit - Much improved | 2 | 2
  Visit 6 Clinic Efficacy Visit - Minimally improved | 3 | 0
  Visit 6 Clinic Efficacy Visit - No change | 9 | 4
  Visit 6 Clinic Efficacy Visit - Minimally worse | 1 | 1
  Visit 7 Clinic Efficacy Visit - Very much improved | 1 | 0
  Visit 7 Clinic Efficacy Visit - Much improved | 4 | 1
  Visit 7 Clinic Efficacy Visit - Minimally improved | 3 | 1
  Visit 7 Clinic Efficacy Visit - No change | 6 | 5
  Visit 7 Clinic Efficacy Visit - Minimally worse | 1 | 0

14. Secondary Outcome: Change From Baseline in Dyskinesia Scores Measured by the Kinesia 360 (Great Lakes Neurotechnologies, Inc) Wearable Dyskinesia Assessment System - Absolute Change From Baseline
Description: The Kinesia 360 (Great Lakes Neurotechnologies, Inc) wearable dyskinesia assessment system was used to monitor dyskinesias. Sensors worn on the wrist and ankle combined with a mobile application continuously record data for assessment dyskinesia. Algorithms were used to detect symptoms from the motion sensors data and calculate a severity score (0 to 1 where score 0 corresponds to no dyskinesia and score 1 corresponds to dyskinesia) every 2 minutes. Wearable data collection of dyskinesia took place during a 2-day period prior to Visit 2 (Baseline), Visit 6 (Titration) and Visit 7 (Steady state). Outcome is presented as the mean ratio at baseline and absolute ratio change from baseline.
Time Frame: Baseline - prior to Day 1 (Visit 2), Titration - prior to Day 28 (Visit 6), and Steady state prior to Day 42 (Visit 7).
Population: Per protocol analysis set (one patient excluded in placebo arm due to major protocol deviation).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NLX-112 | Placebo
Number analyzed (Participants) | 15 | 7
score on a scale
  Baseline | 0.1807 (0.1955) | 0.2855 (0.3322)
  Titration: number analyzed (Participants) | 8 | 3
  Titration | -0.06517 (0.06722) | -0.009172 (0.1353)
  Steady-State: number analyzed (Participants) | 6 | 3
  Steady-State | -0.009327 (0.1243) | -0.01630 (0.3166)

ADVERSE EVENTS:
Time Frame: AEs (including SAEs) were collected from the start of IMP administration (Visit 2) until the end-of-study visit (Visit 9), approximately 70 days.
Description: The grading of the severity/intensity (grade 1 to grade 5) of AEs followed the common terminology criteria for AEs (CTCAE) v5.0 [24]. AEs were assessed as unlikely, possibly or probably related to the IMP
Arm/Group | NLX-112 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/9
Other Adverse Events (participants affected / at risk) | 16/18 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NLX-112 (N=18) | Placebo (N=9)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NLX-112 (N=18) | Placebo (N=9)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Dyskinesia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 2 (3)
On and off phenomenon (Nervous system disorders) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 3 (3) | 3 (7)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dissociation (Psychiatric disorders) | 2 (2) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Illusion (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Rapid eye movement sleep behavior disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1)
Systolic hypertension (Vascular disorders) | 1 (1) | 0 (0)
Binocular eye movement disorder (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Erythema of eyelid (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Swelling of eyelid (Eye disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Product communication issue (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Inflammatory marker increased (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT05148884/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT05148884/SAP_002.pdf